CLINICAL TRIAL: NCT03017703
Title: The Role of Aldosterone in Diabetes Related Vascular Disease, a New Therapeutic Target?
Brief Title: The Role of Aldosterone in Circulatory Disorders Within Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Stefan Mortensen, Associate Professor, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H- 15007940
Record Dates: First submitted 2017-01-02; First posted 2017-01-11 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Endothelial Dysfunction; Insulin Resistance
Keywords: Endothelial dysfunction; Insulin resistance; Type 2 diabetes; Mineralocorticoid blocker
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Type 2 Diabetes (Experimental): 8 weeks of treatment with Aldosterone blocker Eplerenone
  Interventions: Drug: Eplerenone
- Healthy (Experimental): 8 weeks of treatment with Aldosterone blocker Eplerenone
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone

SUMMARY:
The importance of Aldosterone for endothelial function and Insulin resistance observed within patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed diabetic < 5 Yrs.
* BMI < 32 kg/m2
* Non-smoking
* Blood pressure < 140/90 mmHg (treatment with maximum of two antihypertensive drugs)

Exclusion Criteria:

* Insulin treatment
* Hypertension (>140/90 mmHg)
* Sequelae to diabetes
* Smoking
* Known chronic diseases
* Pregnancy or birth within 3 month
* Alcohol misuse

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Vascular function | 8 weeks
  Femoral arterial blood flow in response to femoral arterially infused ACh
Insulin sensitivity measured by a insulin clamp | 8 weeks
  Glucose infusion rate during euglycaemic-hyperinsulinaemic clamp

SECONDARY OUTCOMES:
Vascular function | 8 weeks
  Microperfusion performed on blood vessels in vitro obtained from muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Stefan P Mortensen, DMSc, Principal Investigator — University of Southern Denmark
Locations (1):
- Cardiovascular and Renal Research, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finsen SH, Hansen MR, Hoffmann-Petersen J, Hojgaard HF, Mortensen SP. Eight weeks of mineralocorticoid blockade does not improve insulin sensitivity in type 2 diabetes. Physiol Rep. 2021 Aug;9(15):e14971. doi: 10.14814/phy2.14971. PMID 34350730
- [Derived] Finsen SH, Hansen MR, Hansen PBL, Mortensen SP. Aldosterone Induces Vasoconstriction in Individuals with Type 2 Diabetes: Effect of Acute Antioxidant Administration. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1262-e1270. doi: 10.1210/clinem/dgaa867. PMID 33247722